CLINICAL TRIAL: NCT04904887
Title: Clinical Outcomes With a New Monofocal Intraocular Lens Enhanced for Intermediate Vision
Brief Title: Clinical Outcomes With a New Monofocal IOL Enhanced for Intermediate Vision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dar Al Shifa Hospital (Other)
Responsible Party: Principal Investigator, magda torky, catract and refractive surgery specialist, Dar Al Shifa Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02282021065725
Record Dates: First submitted 2021-05-21; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia | interventions — Phacoemulsification

STUDY DESIGN:
Intervention Model Description: patients undergoing cataract surgery are managed with phacoemulsification and insertion of Eyehance intraocular lens in order to improve their intermediate vision.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessment of intermediate vision, defocus curve (Other): Standardized logarithm of the minimum angle of resolution (logMAR) charts were used for visual acuity measurement at 4 m, 80 cm, and 40 cm.
  he binocular defocus curve: The binocular defocus curve was done to evaluate the functional range of vision. The curve was obtained while the patient wearing his distance correction to provide the best distance visual acuity in both eyes. The test was performed under photopic conditions (85 candelas/m2) using ETDRS charts at a distance of 4m with the introduction of defocusing lenses from +1.00 D to -4.00 D in 0.50 D steps.
  Interventions: Procedure: phacoemulsification

INTERVENTIONS:
Procedure: phacoemulsification — phacoemulsification with implantation of EYEHANCE IOL

SUMMARY:
phacoemulsification with insertion of EYHANCE IOL to improve near and intermediate vision

DETAILED DESCRIPTION:
insertion of new intraocular lens enhanced for intermediate vision

ELIGIBILITY:
Inclusion Criteria:

* normal ocular examination apart from cataract.

Exclusion Criteria:

* previous ocular surgery.
* ocular pathology or corneal abnormalities.
* endothelial cell count below 2000 cells/mm2.
* corneal astigmatism greater than 1.0 diopter (D) measured with Scheimpflug tomography (Sirius, CSO, Italy).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
intermediate vision assessment | 6 months postoperatively
  Standardized logarithm of the minimum angle of resolution (logMAR) charts were used for visual acuity measurement at 80 cm .
near vision assessment | 6 months postoperatively
  Standardized logarithm of the minimum angle of resolution (logMAR) charts were used for visual acuity measurement at 40 cm.

SECONDARY OUTCOMES:
defocus curve | 6 months postoperatively
  The curve was obtained while the patient wearing his distance correction to provide the best distance visual acuity in both eyes. The test was performed under photopic conditions (85 candelas/m2) using ETDRS charts at a distance of 4m with the introduction of defocusing lenses from +1.00 D to -4.00 D in 0.50 D steps.

CONTACTS AND LOCATIONS:
Locations (1):
- Daralshifa hospital, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No